CLINICAL TRIAL: NCT04751474
Title: The Effect of Motivational Messages on Optimism, Hopelessness and Life Satisfaction of Intensive Care Nurses During the COVID-19 Pandemic : A Randomized Controlled Study
Brief Title: The Effect of Motivational Messages on Optimism, Hopelessness and Life Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Elif Gezginci, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2021/47-31
Record Dates: First submitted 2021-02-08; First posted 2021-02-12 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Motivation; Optimism; Hopelessness; Life Satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational messages (Experimental): Participants in the motivational group were sent to motivational messages to their mobile phones for 21 days.
  Interventions: Other: Motivational messages
- Control group (No Intervention): The control group did not receive any intervention.

INTERVENTIONS:
Other: Motivational messages — Participants in the motivational group were sent to motivational messages to their mobile phones for 21 days.
  Arms: Motivational messages

SUMMARY:
The Covid-19 pandemic has affected global health systems and required healthcare professionals to show high performance. In this process, the mental health of intensive care nurses, who undertake the biggest burden in health systems, is negatively affected by the high working hours and patient care burden during the pandemic. When the literature is reviewed, pessimistic thinking, feeling hopeless and not enjoying life at more exacerbated levels can be observed in intensive care nurses. It is concluded that studies are needed to increase the motivation of intensive care nurses during the Covid-19 pandemic.In this study, it was aimed to evaluate the effect of motivational messages on optimism, hopelessness and life satisfaction of intensive care nurses during the Covid-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* agreeing to participate in the study
* being a nurse
* working in intensive care during the COVID-19 pandemic

Exclusion Criteria:

* underfilling or not fill out forms and scales

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Optimistic level assessed by the Life Orientation Test | 21 days after from baseline
  The primary endpoint of this study was the difference between groups in terms of Life Orientation Test scores 21 days after. The scale consists of a total of 10 items. The range of scores obtained from the scale varies between 6-30 points. Low scores indicate pessimism, while high scores indicate optimism.
Hopelessness level assessed by the Beck Hopelessness Scale | 21 days after from baseline
  The primary endpoint of this study was the difference between groups in terms of Beck Hopelessness Scale scores 21 days after. The scale consists of a total of 20 items..The range of scores obtained from the scale varies between 0-20 points. High scores indicate that the level of hopelessness is also high.
Life satisfaction assessed by the Satisfaction with Life Scale | 21 days after from baseline
  The primary endpoint of this study was the difference between groups in terms of Satisfaction with Life Scale scores 21 days after. The scale consists of a total of 5 items.The range of scores obtained from the scale varies between 5-25 points. As the total score obtained from the scale increases, life satisfaction level also increases.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Gezginci, RN, PhD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Elif Gezginci, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shen X, Zou X, Zhong X, Yan J, Li L. Psychological stress of ICU nurses in the time of COVID-19. Crit Care. 2020 May 6;24(1):200. doi: 10.1186/s13054-020-02926-2. No abstract available. PMID 32375848
- [Background] Azoulay E, Cariou A, Bruneel F, Demoule A, Kouatchet A, Reuter D, Souppart V, Combes A, Klouche K, Argaud L, Barbier F, Jourdain M, Reignier J, Papazian L, Guidet B, Geri G, Resche-Rigon M, Guisset O, Labbe V, Megarbane B, Van Der Meersch G, Guitton C, Friedman D, Pochard F, Darmon M, Kentish-Barnes N. Symptoms of Anxiety, Depression, and Peritraumatic Dissociation in Critical Care Clinicians Managing Patients with COVID-19. A Cross-Sectional Study. Am J Respir Crit Care Med. 2020 Nov 15;202(10):1388-1398. doi: 10.1164/rccm.202006-2568OC. PMID 32866409
- [Background] Shechter A, Diaz F, Moise N, Anstey DE, Ye S, Agarwal S, Birk JL, Brodie D, Cannone DE, Chang B, Claassen J, Cornelius T, Derby L, Dong M, Givens RC, Hochman B, Homma S, Kronish IM, Lee SAJ, Manzano W, Mayer LES, McMurry CL, Moitra V, Pham P, Rabbani L, Rivera RR, Schwartz A, Schwartz JE, Shapiro PA, Shaw K, Sullivan AM, Vose C, Wasson L, Edmondson D, Abdalla M. Psychological distress, coping behaviors, and preferences for support among New York healthcare workers during the COVID-19 pandemic. Gen Hosp Psychiatry. 2020 Sep-Oct;66:1-8. doi: 10.1016/j.genhosppsych.2020.06.007. Epub 2020 Jun 16. PMID 32590254
- [Background] Murat M, Kose S, Savaser S. Determination of stress, depression and burnout levels of front-line nurses during the COVID-19 pandemic. Int J Ment Health Nurs. 2021 Apr;30(2):533-543. doi: 10.1111/inm.12818. Epub 2020 Nov 21. PMID 33222350
- [Background] Chen Q, Liang M, Li Y, Guo J, Fei D, Wang L, He L, Sheng C, Cai Y, Li X, Wang J, Zhang Z. Mental health care for medical staff in China during the COVID-19 outbreak. Lancet Psychiatry. 2020 Apr;7(4):e15-e16. doi: 10.1016/S2215-0366(20)30078-X. Epub 2020 Feb 19. No abstract available. PMID 32085839
- [Background] Lissoni B, Del Negro S, Brioschi P, Casella G, Fontana I, Bruni C, Lamiani G. Promoting resilience in the acute phase of the COVID-19 pandemic: Psychological interventions for intensive care unit (ICU) clinicians and family members. Psychol Trauma. 2020 Aug;12(S1):S105-S107. doi: 10.1037/tra0000802. Epub 2020 Jun 18. PMID 32551763
- [Background] Schulte EE, Bernstein CA, Cabana MD. Addressing Faculty Emotional Responses during the Coronavirus 2019 Pandemic. J Pediatr. 2020 Jul;222:13-14. doi: 10.1016/j.jpeds.2020.04.057. Epub 2020 May 7. No abstract available. PMID 32387715
- [Background] Chung JPY, Yeung WS. Staff Mental Health Self-Assessment During the COVID-19 Outbreak. East Asian Arch Psychiatry. 2020 Mar;30(1):34. doi: 10.12809/eaap2014. No abstract available. PMID 32229646
- [Derived] Kose S, Gezginci E, Goktas S, Murat M. The effectiveness of motivational messages to intensive care unit nurses during the COVID-19 pandemic. Intensive Crit Care Nurs. 2022 Apr;69:103161. doi: 10.1016/j.iccn.2021.103161. Epub 2021 Nov 1. PMID 34895798